CLINICAL TRIAL: NCT01946646
Title: A Phase I Study of TS-1 With Concurrent Radiotherapy Followed by Gemcitabine and TS-1 in Metastatic Pancreatic Cancer (SR-GS Study)
Brief Title: Phase I Study of TS-1 With Concurrent Radiotherapy to Treat Pancreatic Cancer
Acronym: SR-GS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: National Taiwan University Hospital (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201211048MPC
Record Dates: First submitted 2013-09-11; First posted 2013-09-19 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1-CCRT (Experimental): There are five dose levels and one arm only. Level 1: S-1, 25 mg/m2, bid, Day 1-14; RT 25 Gy/10 fx, Day 1-5, 8-12 Level 2: S-1, 25 mg/m2, bid, Day 1-14; RT 30 Gy/10 fx, Day 1-5, 8-12 Level 3: S-1, 30 mg/m2, bid, Day 1-14; RT 30 Gy/10 fx, Day 1-5, 8-12 Level 4: S-1, 30 mg/m2, bid, Day 1-16; RT 36 Gy/12 fx, Day 1-5, 8-12, 15-16 Level 5: S-1, 35 mg/m2, bid, Day 1-16; RT 36 Gy/12 fx, Day 1-5, 8-12, 15-16 All dose levels are followed by Gemcitabine/S-1 (G 1000 mg/m2, iv, D1 and 15 plus S-1 60/80/100 mg/day based on BSA, po, D1-7, D15-21, q4w) after the CCRT
  Interventions: Drug: S-1-CCRT

INTERVENTIONS:
Drug: S-1-CCRT

SUMMARY:
The purpose of this study is to determine whether combination of TS-1 and concurrent and short-course radiotherapy is feasible in metastatic pancreatic cancer. The rationale of this study primarily bases on the good efficacy of gemcitabine plus TS-1 and the great potential of local control of concurrent chemoradiotherapy in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven, newly diagnosed pancreatic adenocarcinoma or adenosquamous carcinoma
* no previous radiotherapy, chemotherapy, targeted therapy, curative surgery, or immunotherapy used for pancreatic cancer
* presence of at least one measurable lesion, which must meet the criteria of being ≥ 20 mm in at least one dimension by conventional CT/MRI or ≥ 10 mm by spiral CT scan
* age between 20 and 79 years at registration
* ECOG PS of 0 or 1
* adequate major organ functions
* ability to take the oral study medication (TS-1)
* no clinically significant abnormal ECG findings within 28 days (4 weeks) prior to registration
* voluntarily signed the written informed consent form

Exclusion Criteria:

* pulmonary fibrosis or interstitial pneumonitis diagnosed within 28 days prior to registration
* presence of diarrhea ≥ CTCAE v.4.03 grade 2
* concomitant active infection or significant co-morbid medical conditions
* moderate or severe ascites or pleural effusion that requires drainage
* central nervous system metastasis
* prior or concurrent malignancies within the last 3 years
* concomitant treatment with flucytosine, phenytoin or warfarin
* pregnant women or nursing mothers, or positive pregnancy test
* severe mental disorder
* judged ineligible by physician for participation in the study due to safety concern

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 weeks
  Dose-limiting toxicities (DLT) are defined as the following manifestations of toxicity observed until completion of CCRT:
  1. grade 3 leucopenia and/or neutropenia with a fever ≥ 38°C lasting 3 days or more
  2. grade 3 leucopenia and/or neutropenia with infection
  3. grade 4 leucopenia and/or neutropenia lasting 3 days or more
  4. grade 4 leucopenia and/or neutropenia requiring G-CSF
  5. platelet < 25,000/mm3
  6. , grade 3 thrombocytopenia requiring transfusion
  7. hemoglobin < 8.0 g/dL
  g. serum AST/ALT ≥ 10 times ULN h. total bilirubin ≥ 3 times ULN i. creatinine >3.0 - 6.0 times ULN (grade 3) i. grade 3 or 4 nonhematological toxicities including nausea, vomiting, anorexia, fatigue, constipation, hyperglycemia, and abnormality of sodium, potassium, and calcium If three or more patients experience DLT at a given dose level, then the previous dose level will be considered as the MTD.
maximum-tolerated dose | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan